CLINICAL TRIAL: NCT02850731
Title: Motorized Platform and Autonomy Among the Frail and Pre-frail Older Adult
Brief Title: Motorized Platform and Autonomy Among the Frail and Pre-frail Older Adult (PLATAUTONOMIE)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisation problem
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15 7841 16
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Fragility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plate-forme Hu360® (Experimental): the innovative technology (plate-forme Hu360®) will be used in the experimental arm
  Interventions: Device: plate-forme Hu360®
- supervision by a therapist (No Intervention): an adapted physical activity program under supervision of a therapist

INTERVENTIONS:
Device: plate-forme Hu360® — the innovative technology (plate-forme Hu360®) will be used in the experimental arm
  Arms: plate-forme Hu360®

SUMMARY:
Highly diversified programs of physical activity in older people have shown their effectiveness in terms of improving functional capacities. Only one of these programs, to date, has used a motorized platform. The motorized platform allows the use of sensorimotor programs adapted to this population. Thus, for the user, a combination of motor and sensory capacities necessary to actively control different positions as well as reactions to maintain balance are stimulated, and are as important as psychomotor capabilities to maintain autonomy and the fight against losing independence.

Demonstration of the effectiveness of this type of equipment would propose a new modality of physical activity adapted to this population. Use of this new equipment could allow the possibility of standardizing this activity, whilst continuing to individualize physical activity programs.

Two phases for each group (Intervention/Control):

Phase 1 (day 0 - week 6): 2x1 hour sessions per week using the Hu360® (Intervention group) or an adapted physical activity program (Control group) under supervision of a therapist who will adapt the program according to the progress of the patient, following a standardized procedure (exercises: postural/balance training, strength training for the legs/trunk and coordination and endurance activities) Phase 2 (week 6 - month 6): Physical activity program at home for both groups, performed independently.

Blinded evaluations will be performed at 6 weeks and at 6 months for each group.

The investigators hypothesis is that the use of the motorized platform will allow superior physical performance compared to a traditional physical activity program.

DETAILED DESCRIPTION:
Background

The process of aging causes a progressive decline in functional capacities. Maintaining physical fitness appears to be an important factor to fight against frailty (40% more frailty in people > 65 years old), a condition that causes loss of independence but that is clinically reversible.

Fragility is a condition that associates: slowed walking speed, sedentary lifestyle, weight loss, muscle weakness and low energy levels. It is therefore correlated with physical performance.

Purpose

A number of studies have demonstrated the benefit of physical activity in frail older people. Levels of adherence to physical activity programs are not well known but low adherence decreases the positive effects of the intervention. It seems therefore interesting to suggest another approach that integrates innovative technology (plate-forme Hu360®) that can improve the clinical condition of the frail older person, as well as levels of adherence.

Abstract

Highly diversified programs of physical activity in older people have shown their effectiveness in terms of improving functional capacities. Only one of these programs, to date, has used a motorized platform. The motorized platform allows the use of sensorimotor programs adapted to this population. Thus, for the user, a combination of motor and sensory capacities necessary to actively control different positions as well as reactions to maintain balance are stimulated, and are as important as psychomotor capabilities to maintain autonomy and the fight against losing independence.

Demonstration of the effectiveness of this type of equipment would propose a new modality of physical activity adapted to this population. Use of this new equipment could allow the possibility of standardizing this activity, whilst continuing to individualize physical activity programs.

Two phases for each group (Intervention/Control):

Phase 1 (day 0 - week 6): 2x1 hour sessions per week using the Hu360® (Intervention group) or an adapted physical activity program (Control group) under supervision of a therapist who will adapt the program according to the progress of the patient, following a standardized procedure (exercises: postural/balance training, strength training for the legs/trunk and coordination and endurance activities)

Phase 2 (week 6 - month 6): Physical activity program at home for both groups, performed independently.

Blinded evaluations will be performed at 6 weeks and at 6 months for each group.

The investigators hypothesis is that the use of the motorized platform will allow superior physical performance compared to a traditional physical activity program.

Statistical analysis

Data analysis will be realized, blinded to the treatment group. The analysis will be conducted with intention to treat.

The principal analysis will be made using a linear mixed model for repeated data, taking into account stratification factors (gender and class Score SPPB at baseline) by random effect, without imputation of missing data. An exploratory analysis will be conducted on the principal outcome measure using a linear mixed model for repeated data, taking into account stratification factors and some covariates that may change the effect of the intervention, such compliance.

Secondary outcome measures will be will be analysed in a similar manner by generalized linear mixed models. The tests will be bilateral. An error-correction modem of 5% will be considered during the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 70-89 years old.
* Living at home
* Having at least one fragility criteria (from Fried's 5 criteria), which must include the sedentary criteria.
* Having a Score SPPB <10
* Independent mobility
* MMSE score ≥18
* BMI between 18 and 40
* Informed consent to participate in a randomized control trial (physical activity using the motorized platform, Hu360® vs a traditional physical activity program).

Exclusion Criteria:

* Severe cardiac problems
* Degenerative neurological conditions
* Hip/Knee joint replacement less than 6 months before the study.
* Psychotic disorders or bipolar disorder.
* Patients who already participate in a regular physical activity program or follow a rehabilitation program.
* Patients under legal protection and / or unable to give informed consent
* Already participating in a clinical trial or a study with a physical activity program.

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of physical performances using the Score Short Physical Performance Battery | 6 months
  Evolution of physical performances within 6 months estimated by the Score Short Physical Performance Battery

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Carette, PhD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No